CLINICAL TRIAL: NCT01986933
Title: A PHASE II, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, MULTIPLE-DOSE STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND EFFICACY OF CIM331 IN ATOPIC DERMATITIS PATIENTS WHO ARE INADEQUATELY CONTROLLED BY OR INTOLERANT TO TOPICAL THERAPY
Brief Title: A Phase 2 Study of CIM331 for Atopic Dermatitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIM003JG
Record Dates: First submitted 2013-10-31; First posted 2013-11-19 (Estimated); Results first posted 2021-11-22 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — nemolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group1 (Experimental): Part A: nemolizumab (CIM331) Part B: nemolizumab (CIM331)
  Interventions: Drug: nemolizumab (CIM331)
- Group2 (Experimental): Part A: nemolizumab (CIM331) Part B: nemolizumab (CIM331)
  Interventions: Drug: nemolizumab (CIM331)
- Group3 (Experimental): Part A: nemolizumab (CIM331) Part B: nemolizumab (CIM331)
  Interventions: Drug: nemolizumab (CIM331)
- Group4 (Experimental): Part A: nemolizumab (CIM331) Part B: nemolizumab (CIM331)
  Interventions: Drug: nemolizumab (CIM331)
- Group5 (Experimental): Part A: Placebo Part B: nemolizumab (CIM331)
  Interventions: Drug: nemolizumab (CIM331); Other: Placebo

INTERVENTIONS:
Drug: nemolizumab (CIM331)
Other: Placebo
  Arms: Group5

SUMMARY:
To assess the safety, tolerability and efficacy of CIM331, compared to placebo, in atopic dermatitis patients who are inadequately controlled by or intolerant to topical therapy

ELIGIBILITY:
Inclusion Criteria:

* ≥18 and ≤65 years of age at the time of consent.
* Patients with Atopic Dermatitis
* Pruritus visual analogue scale (VAS) ≥50 mm at the screening and baseline visit
* Eczema Area and Severity Index (EASI) ≥10 at the screening and baseline visit
* static Investigator's Global Assessment (sIGA) score ≥3 at the baseline visit

Exclusion Criteria:

* Serological evidence of hepatitis B virus or hepatitis C virus infection
* Known human immunodeficiency virus infection
* Ongoing treatment with specific or non-specific hyposensitization therapy for AD
* Treatment with mild or moderately potent topical corticosteroids (TCS) within 1 week prior to randomization
* History of infection including skin infection requiring treatment with oral or intravenous (IV) antibiotics, antivirals, or antifungals within 1 week prior to randomization.
* Evidence of tuberculosis (TB) infection as defined by a positive purified protein derivative (PPD) and/or positive interferon-gamma release assay.
* Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2013-11; Primary Completion 2015-04 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryosuke Mihara, Study Director — Chugai Pharmaceutical
Locations (16):
- United States (16):
  - Anniston, Alabama
  - San Diego, California
  - Miami, Florida
  - Alpharetta, Georgia
  - Arlington Heights, Illinois
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Bay City, Michigan
  - New York, New York
  - Charlotte, North Carolina
  - Cleveland, Ohio
  - Portland, Oregon
  - Charleston, South Carolina
  - College Station, Texas
  - Norfolk, Virginia

REFERENCES:
- [Derived] Kabashima K, Furue M, Hanifin JM, Pulka G, Wollenberg A, Galus R, Etoh T, Mihara R, Nakano M, Ruzicka T. Nemolizumab in patients with moderate-to-severe atopic dermatitis: Randomized, phase II, long-term extension study. J Allergy Clin Immunol. 2018 Oct;142(4):1121-1130.e7. doi: 10.1016/j.jaci.2018.03.018. Epub 2018 May 10. PMID 29753033
- [Derived] Ruzicka T, Hanifin JM, Furue M, Pulka G, Mlynarczyk I, Wollenberg A, Galus R, Etoh T, Mihara R, Yoshida H, Stewart J, Kabashima K; XCIMA Study Group. Anti-Interleukin-31 Receptor A Antibody for Atopic Dermatitis. N Engl J Med. 2017 Mar 2;376(9):826-835. doi: 10.1056/NEJMoa1606490. PMID 28249150

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were enrolled at 57 investigational sites in the UK, Germany, Poland, Japan, and the US.
Pre-assignment Details: Patient eligibility was assessed during the screening period (Day -28 to Day -8). If all eligibility criteria were met, the patient entered a 7-day run-in period (Day -7 to Day -1) during which all prohibited treatments were discontinued. Baseline assessments were performed until randomization on Day 1.
Groups:
- Placebo: The study was undertaken in two parts, Part A and Part B. A Safety Follow-up visit was performed 12 weeks after the last dose of study drug.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received placebo subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
  Placebo-to-active period (Part B ) (up to Week 64):
  Patients randomized to placebo group in Part A were re-randomized to Nemoliozumab groups (0.1 mg/kg, 0.5 mg/kg or 2.0 mg/kg Q4W) in Part B. Nemoliozumab was given subcutaneously every 4 weeks for 52 weeks. Placebo-treated patients in Part A were not re-randomized to Nemoliozumab (2.0 mg/kg) Q8W group in Part B.
- Nemoliozumab (0.1 mg/kg) Q4W: The study was undertaken in two parts, Part A and Part B. A Safety Follow-up visit was performed 12 weeks after the last dose of study drug.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (0.1 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
  Active-to-active period (Part B ) (up to Week 64):
  Patients in the Nemoliozumab (0.1 mg/kg) Q4W group during Part A continuously used the same regimen of Nemoliozumab in Part B.
  Placebo-to-active period (Part B) (up to Week 64):
  Patients in the Placebo group during Part A were re-randomized to Nemoliozumab groups (0.1 mg/kg, 0.5 mg/kg or 2.0 mg/kg Q4W) in Part B.
- Nemoliozumab (0.5 mg/kg) Q4W: The study was undertaken in two parts, Part A and Part B. A Safety Follow-up visit was performed 12 weeks after the last dose of study drug.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (0.5 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
  Active-to-active period (Part B ) (up to Week 64):
  Patients in the Nemoliozumab (0.5 mg/kg) Q4W group during Part A continuously used the same regimen of Nemoliozumab in Part B.
  Placebo-to-active period (Part B) (up to Week 64):
  Patients in the Placebo group during Part A were re-randomized to Nemoliozumab groups (0.1 mg/kg, 0.5 mg/kg or 2.0 mg/kg Q4W) in Part B.
- Nemoliozumab (2.0 mg/kg) Q4W: The study was undertaken in two parts, Part A and Part B. A Safety Follow-up visit was performed 12 weeks after the last dose of study drug.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (2.0 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
  Active-to-active period (Part B ) (up to Week 64):
  Patients in the Nemoliozumab (2.0 mg/kg) Q4W group during Part A continuously used the same regimen of Nemoliozumab in Part B.
  Placebo-to-active period (Part B) (up to Week 64):
  Patients in the Placebo group during Part A were re-randomized to Nemoliozumab groups (0.1 mg/kg, 0.5 mg/kg or 2.0 mg/kg Q4W) in Part B.
- Nemoliozumab (2.0 mg/kg) Q8W: The study was undertaken in two parts, Part A and Part B. A Safety Follow-up visit was performed 12 weeks after the last dose of study drug.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (2.0 mg/kg) subcutaneously every 8 weeks on Day 1 and Week 8.
  Active-to-active period (Part B ) (up to Week 64):
  Patients in the Nemoliozumab (2.0 mg/kg) Q8W group during Part A continuously used the same regimen of Nemoliozumab in Part B.
  Placebo-to-active period (Part B) (up to Week 64):
  Placebo-treated patients in Part A were not re-randomized to Nemoliozumab (2.0 mg/kg) Q8W group in Part B.
Period: Placebo-controlled (Part A)
Arm/Group | Placebo | Nemoliozumab (0.1 mg/kg) Q4W | Nemoliozumab (0.5 mg/kg) Q4W | Nemoliozumab (2.0 mg/kg) Q4W | Nemoliozumab (2.0 mg/kg) Q8W
Started (Patients were randomly assigned (1:1:1:1:1 ratio) to one of four active treatment groups and one placebo group in double-blind fashion.) | 53 | 53 | 54 | 52 | 52
Completed | 44 | 44 | 45 | 45 | 38
Not Completed | 9 | 9 | 9 | 7 | 14
Not completed — Adverse Event | 1 | 5 | 2 | 2 | 4
Not completed — Lack of Efficacy | 3 | 1 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 5 | 2 | 6 | 2 | 7
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0
Not completed — Others (not classified above reasons) | 0 | 0 | 0 | 0 | 2
Period: Active-to-active (Part B)
Arm/Group | Placebo | Nemoliozumab (0.1 mg/kg) Q4W | Nemoliozumab (0.5 mg/kg) Q4W | Nemoliozumab (2.0 mg/kg) Q4W | Nemoliozumab (2.0 mg/kg) Q8W
Started (Data from patients who were randomized to Nemoliozumab groups in Part A and initiated Part B were analyzed.) | 0 | 41 | 38 | 39 | 35
Completed | 0 | 31 | 28 | 30 | 19
Not Completed | 0 | 10 | 10 | 9 | 16
Not completed — Adverse Event | 0 | 2 | 0 | 1 | 3
Not completed — Lack of Efficacy | 0 | 3 | 2 | 0 | 4
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 7 | 6 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Others (not classified above reasons) | 0 | 1 | 0 | 1 | 1
Period: Placebo-to-active (Part B)
Arm/Group | Placebo | Nemoliozumab (0.1 mg/kg) Q4W | Nemoliozumab (0.5 mg/kg) Q4W | Nemoliozumab (2.0 mg/kg) Q4W | Nemoliozumab (2.0 mg/kg) Q8W
Started (Data from patients who were randomized to placebo group in Part A and initiated Part B were analyzed.) | 0 | 13 (Patients in the initial placebo group were re-randomized into Nemoliozumab groups (0.1, 0.5 or 2.0 mg/kg Q4W) in Part B.) | 12 (Patients in the initial placebo group were re-randomized into Nemoliozumab groups (0.1, 0.5 or 2.0 mg/kg Q4W) in Part B.) | 13 (Patients in the initial placebo group were re-randomized into Nemoliozumab groups (0.1, 0.5 or 2.0 mg/kg Q4W) in Part B.) | 0 (Patients in the initial placebo group were not re-randomized into Nemoliozumab (2.0 mg/kg) Q8W group in Part B.)
Completed | 0 | 8 | 7 | 8 | 0
Not Completed | 0 | 5 | 5 | 5 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 4 | 3 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The per-protocol (PP) population in Part A was used for the analysis. The PP population was defined as a subset of the intent to treat (ITT) population excluding some of the major protocol violators, patients who were withdrawn before being evaluated for pruritus Visual Analogue Scale (VAS) at Week 8, or those who withdrew prior to receiving two or more study drug administrations. Patients who received the wrong study drug were also excluded from the PP population.
Groups:
- Placebo (Part A): Data from patients randomized to this group in Part A were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received placebo subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
- Nemoliozumab (0.1 mg/kg) Q4W (Part A): Data from patients randomized to this group in Part A were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (0.1 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
- Nemoliozumab (0.5 mg/kg) Q4W (Part A): Data from patients randomized to this group in Part A were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (0.5 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
- Nemoliozumab (2.0 mg/kg) Q4W (Part A): Data from patients randomized to this group in Part A were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (2.0 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
- Nemoliozumab (2.0 mg/kg) Q8W (Part A): Data from patients randomized to this group in Part A were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (2.0 mg/kg) subcutaneously every 8 weeks on Day 1 and Week 8.
- Total: Total of all reporting groups
Arm/Group | Placebo (Part A) | Nemoliozumab (0.1 mg/kg) Q4W (Part A) | Nemoliozumab (0.5 mg/kg) Q4W (Part A) | Nemoliozumab (2.0 mg/kg) Q4W (Part A) | Nemoliozumab (2.0 mg/kg) Q8W (Part A) | Total
Number analyzed (Participants) | 46 | 46 | 45 | 47 | 45 | 229
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (13.3) | 33.9 (10.2) | 33.0 (11.5) | 33.7 (12.2) | 34.6 (13.3) | 34.2 (12.1)
Age, Customized [Count of Participants; unit: Participants]
  Age Category: < 20 years | 4 | 0 | 3 | 1 | 1 | 9
  Age Category: 20 -< 30 years | 14 | 21 | 22 | 20 | 21 | 98
  Age Category: 30 -< 40 years | 10 | 15 | 7 | 13 | 7 | 52
  Age Category: 40 -< 50 years | 8 | 4 | 6 | 7 | 7 | 32
  Age Category: 50 -< 60 years | 8 | 6 | 7 | 4 | 7 | 32
  Age Category: > 60 years | 2 | 0 | 0 | 2 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 27 | 18 | 21 | 110
  Male | 23 | 25 | 18 | 29 | 24 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 45 | 45 | 44 | 45 | 44 | 223
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 13 | 17 | 11 | 15 | 14 | 70
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 6 | 1 | 4 | 15
  White | 32 | 26 | 27 | 30 | 27 | 142
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Height [Mean (Standard Deviation); unit: Centimetre] | 167.81 (8.84) | 170.19 (10.52) | 167.41 (9.44) | 170.04 (8.84) | 167.58 (9.63) | 168.62 (9.47)
Weight [Mean (Standard Deviation); unit: Kilogram] | 74.20 (21.60) | 76.01 (22.90) | 73.40 (19.98) | 72.51 (16.04) | 72.63 (20.96) | 73.75 (20.27)
Weight Category [Count of Participants; unit: Participants]
  < 60 kg | 11 | 12 | 15 | 11 | 15 | 64
  >- 60 kg | 35 | 34 | 30 | 36 | 30 | 165
Body mass index [Mean (Standard Deviation); unit: Kilogram per square metre] | 26.20 (6.81) | 25.92 (6.41) | 26.10 (6.66) | 25.08 (5.26) | 25.71 (6.47) | 25.80 (6.30)
Body Mass Index Category [Count of Participants; unit: Participants]
  < 25 kg/m^2 | 27 | 26 | 23 | 28 | 23 | 127
  >- 25 kg/m^2 | 19 | 20 | 22 | 19 | 22 | 102

OUTCOME MEASURES:

1. Primary Outcome: Percent Changes From Baseline in Pruritus Visual Analogue Scale (VAS) at Week 12
Description: Percent changes from baseline in pruritus VAS at Week 12. VAS indicates pruritus intensity in the last 24 hours, from 0 (no itch) to 10 (worst imaginable itch).
  When condition of pruritus improves, percent change from baseline at Week 12 indicates negative value (i.e. the higher the absolute value is, the more the condition improves).
Time Frame: baseline to Week 12
Population: The per-protocol (PP) population in Part A was used for the analysis. The PP population was defined as a subset of the intent to treat (ITT) population excluding some of the major protocol violators, patients who were withdrawn before being evaluated for pruritus VAS at Week 8, or those who withdrew prior to receiving two or more study drug administrations. Patients who received the wrong study drug were also excluded from the PP population.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage change
Groups:
- Placebo (Part A): Data from Part A were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received placebo subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
- Nemoliozumab (0.1 mg/kg) Q4W (Part A): Data from Part A were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (0.1 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
- Nemoliozumab (0.5 mg/kg) Q4W (Part A): Data from Part A were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (0.5 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
- Nemoliozumab (2.0 mg/kg) Q4W (Part A): Data from Part A were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (2.0 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
Arm/Group | Placebo (Part A) | Nemoliozumab (0.1 mg/kg) Q4W (Part A) | Nemoliozumab (0.5 mg/kg) Q4W (Part A) | Nemoliozumab (2.0 mg/kg) Q4W (Part A)
Number analyzed (Participants) | 43 | 44 | 43 | 46
percentage change | -20.07 [-29.94 to -10.21] | -41.46 [-51.21 to -31.71] | -61.24 [-71.13 to -51.35] | -60.46 [-69.98 to -50.95]
Statistical Analysis 1: Comparison: Placebo (Part A) vs Nemoliozumab (0.1 mg/kg) Q4W (Part A); Test type: Superiority; p = 0.0027, ANCOVA — Since a hierarchical decision procedure can be regarded as a closed testing procedure, no inflation of the alpha level due to multiple comparisons was necessary, and the global 1-sided significance alpha level of 0.025 was maintained; Mean Difference (Final Values) = -21.39, 95% CI 2-sided [-35.25 to -7.53], Standard Error of Mean 7.02
Statistical Analysis 2: Comparison: Placebo (Part A) vs Nemoliozumab (0.5 mg/kg) Q4W (Part A); Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -41.16, 95% CI 2-sided [-55.17 to -27.15], Standard Error of Mean 7.10
Statistical Analysis 3: Comparison: Placebo (Part A) vs Nemoliozumab (2.0 mg/kg) Q4W (Part A); Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -40.39, 95% CI 2-sided [-54.11 to -26.67], Standard Error of Mean 6.95

2. Secondary Outcome: Changes From Baseline in Eczema Area and Severity Index (EASI) (Part A, PP Population)
Description: EASI score was used to measure the severity and extent of atopic eczema. The intensity of a representative area of eczema and the approximate percentage affected by eczema were calculated for each of the four body regions: head and neck, upper limbs, trunk, and lower limbs. The sum of the above 4 body region scores was calculated and should be 0 (none) to 72 (severest).
  When the condition of eczema improves, the percent change from baseline at each timepoint indicates negative value (i.e. the higher the absolute value is, the more the condition improves).
Time Frame: baseline to Week 12 (Part A)
Population: The per-protocol (PP) population in Part A was used for the analysis. The PP population was defined as a subset of the ITT population excluding some of the major protocol violators , patients who were withdrawn before being evaluated for pruritus VAS at Week 8, or those who withdrew prior to receiving two or more study drug administrations. Patients who received the wrong study drug were also excluded from the PP population.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Placebo (Part A) | Nemoliozumab (0.1 mg/kg) Q4W (Part A) | Nemoliozumab (0.5 mg/kg) Q4W (Part A) | Nemoliozumab (2.0 mg/kg) Q4W (Part A)
Number analyzed (Participants) | 46 | 46 | 45 | 47
percentage change from baseline
  Week 4: number analyzed (Participants) | 43 | 44 | 43 | 46
  Week 4 | -12.12 (40.00) | -26.89 (44.48) | -35.70 (44.29) | -33.86 (34.14)
  Week 8: number analyzed (Participants) | 43 | 44 | 43 | 46
  Week 8 | -21.82 (47.00) | -25.17 (51.79) | -46.20 (42.62) | -39.89 (34.43)
  Week 12: number analyzed (Participants) | 43 | 44 | 43 | 46
  Week 12 | -20.89 (47.63) | -27.88 (50.50) | -44.57 (48.21) | -40.29 (37.70)

3. Secondary Outcome: Changes From Baseline in Eczema Area and Severity Index (EASI) (Part A + Part B, ITT Long Population)
Description: as for outcome 2
Time Frame: baseline to Week 12 (Part A), up to Week 64 (Part B)
Population: The intent to treat (ITT) Long population was used for the analysis. The ITT Long population included patients randomized to Nemoliozumab treatment groups in Part A and patients re-randomized from the placebo group to Nemoliozumab treatment groups, providing they received at least one dose of Nemoliozumab and providing the results of at least one post-dose efficacy assessment was available.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Groups:
- Nemoliozumab (0.1 mg/kg) Q4W (Part A + Part B): Data from Part A and Part B were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (0.1 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
  Active-to-active period (Part B) (up to Week 64):
  Patients in the Nemoliozumab (0.1 mg/kg) Q4W group during Part A continuously used the same regimen of Nemoliozumab in Part B.
- Nemoliozumab (0.5 mg/kg) Q4W (Part A + Part B): Data from Part A and Part B were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (0.5 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
  Active-to-active period (Part B) (up to Week 64):
  Patients in the Nemoliozumab (0.5 mg/kg) Q4W group during Part A continuously used the same regimen of Nemoliozumab in Part B.
- Nemoliozumab (2.0 mg/kg) Q4W (Part A + Part B): Data from Part A and Part B were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (2.0 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
  Active-to-active period (Part B) (up to Week 64):
  Patients in the Nemoliozumab (2.0 mg/kg) Q4W group during Part A continuously used the same regimen of Nemoliozumab in Part B.
- Nemoliozumab (2.0 mg/kg) Q8W (Part A + Part B): Data from Part A and Part B were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (2.0 mg/kg) subcutaneously every 8 weeks on Day 1 and Week 8.
  Active-to-active period (Part B) (up to Week 64):
  Patients in the Nemoliozumab (2.0 mg/kg) Q8W group during Part A continuously used the same regimen of Nemoliozumab in Part B.
Arm/Group | Nemoliozumab (0.1 mg/kg) Q4W (Part A + Part B) | Nemoliozumab (0.5 mg/kg) Q4W (Part A + Part B) | Nemoliozumab (2.0 mg/kg) Q4W (Part A + Part B) | Nemoliozumab (2.0 mg/kg) Q8W (Part A + Part B)
Number analyzed (Participants) | 53 | 54 | 52 | 52
percentage change from baseline
  Week 4: number analyzed (Participants) | 51 | 53 | 50 | 46
  Week 4 | -25.47 (42.41) | -32.11 (43.70) | -32.48 (34.02) | -25.43 (35.58)
  Week 8: number analyzed (Participants) | 48 | 45 | 47 | 42
  Week 8 | -25.13 (49.82) | -47.86 (41.38) | -41.02 (36.50) | -33.35 (38.00)
  Week 12: number analyzed (Participants) | 45 | 46 | 46 | 37
  Week 12 | -35.11 (47.92) | -47.75 (45.41) | -46.78 (35.15) | -42.12 (40.82)
  Week 24: number analyzed (Participants) | 38 | 32 | 37 | 29
  Week 24 | -55.83 (42.25) | -62.71 (44.37) | -56.26 (34.68) | -51.01 (37.07)
  Week 48: number analyzed (Participants) | 32 | 29 | 32 | 20
  Week 48 | -69.90 (28.17) | -71.16 (43.31) | -61.14 (44.43) | -74.29 (33.97)
  Week 60: number analyzed (Participants) | 31 | 28 | 32 | 19
  Week 60 | -63.11 (41.89) | -78.81 (28.82) | -70.85 (36.24) | -70.87 (32.84)
  Week 64: number analyzed (Participants) | 31 | 28 | 29 | 19
  Week 64 | -68.45 (41.62) | -75.79 (25.40) | -78.91 (24.34) | -69.25 (43.96)

4. Secondary Outcome: Changes From Baseline in SCORing Atopic Dermatitis (SCORAD) (Part A, PP Population)
Description: SCORAD is a clinical tool used to assess the extent and severity of eczema. Area and intensity, were assessed by the Investigator and subjective symptoms were reported by the patient in order to determine an overall score. The score should be 0 to 103: mild [<25], moderate [25-50] or severe [>50]).
  When the condition of eczema improves, the percent change from baseline at each timepoint indicates negative value (i.e. the higher the absolute value is, the more the condition improves).
Time Frame: baseline to Week 12 (Part A)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Placebo (Part A) | Nemoliozumab (0.1 mg/kg) Q4W (Part A) | Nemoliozumab (0.5 mg/kg) Q4W (Part A) | Nemoliozumab (2.0 mg/kg) Q4W (Part A)
Number analyzed (Participants) | 46 | 46 | 45 | 47
percentage change from baseline
  Week 4: number analyzed (Participants) | 39 | 38 | 39 | 42
  Week 4 | -6.83 (25.97) | -29.31 (23.58) | -34.59 (29.36) | -29.82 (21.65)
  Week 8: number analyzed (Participants) | 39 | 38 | 39 | 42
  Week 8 | -17.29 (30.74) | -26.41 (26.60) | -36.81 (29.04) | -34.72 (24.33)
  Week 12: number analyzed (Participants) | 39 | 38 | 39 | 42
  Week 12 | -15.97 (26.99) | -27.22 (25.81) | -39.49 (32.68) | -38.31 (28.85)

5. Secondary Outcome: Changes From Baseline in SCORing Atopic Dermatitis (SCORAD) (Part A + Part B, ITT Long Population)
Description: as for outcome 4
Time Frame: baseline to Week 12 (Part A), up to Week 64 (Part B)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Nemoliozumab (0.1 mg/kg) Q4W (Part A + Part B) | Nemoliozumab (0.5 mg/kg) Q4W (Part A + Part B) | Nemoliozumab (2.0 mg/kg) Q4W (Part A + Part B) | Nemoliozumab (2.0 mg/kg) Q8W (Part A + Part B)
Number analyzed (Participants) | 53 | 54 | 52 | 52
percentage change from baseline
  Week 4: number analyzed (Participants) | 45 | 47 | 45 | 39
  Week 4 | -27.73 (23.92) | -30.30 (30.39) | -28.20 (22.65) | -25.31 (22.68)
  Week 8: number analyzed (Participants) | 41 | 38 | 41 | 35
  Week 8 | -29.05 (27.17) | -36.16 (28.60) | -37.52 (23.34) | -31.81 (28.42)
  Week 12: number analyzed (Participants) | 39 | 40 | 41 | 32
  Week 12 | -36.35 (22.24) | -42.22 (30.72) | -42.60 (27.12) | -41.85 (20.79)
  Week 24: number analyzed (Participants) | 34 | 27 | 33 | 23
  Week 24 | -48.73 (27.64) | -58.15 (28.15) | -52.00 (24.97) | -49.97 (24.99)
  Week 48: number analyzed (Participants) | 29 | 24 | 29 | 19
  Week 48 | -55.82 (24.21) | -59.20 (28.61) | -53.82 (29.98) | -66.15 (24.43)
  Week 60: number analyzed (Participants) | 28 | 24 | 29 | 18
  Week 60 | -55.08 (24.22) | -64.02 (24.24) | -63.26 (25.04) | -61.03 (24.27)
  Week 64: number analyzed (Participants) | 28 | 23 | 26 | 18
  Week 64 | -56.55 (28.25) | -64.02 (27.72) | -66.61 (19.90) | -63.07 (27.96)

6. Secondary Outcome: Changes From Baseline in Static Investigator's Global Assessment (sIGA) (Part A, PP Population)
Description: The sIGA consisted of a 6-point severity scale from clear to very severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease and 5 = very severe disease). The sIGA assessed clinical characteristics of erythema, infiltration, papulation, oozing and crusting for the overall severity assessment at the time of evaluation.
  When the skin condition improves, the change from baseline at each timepoint indicates negative value (i.e. the higher the absolute value is, the more the condition improves).
Time Frame: baseline to Week 12 (Part A)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: change from baseline
Arm/Group | Placebo (Part A) | Nemoliozumab (0.1 mg/kg) Q4W (Part A) | Nemoliozumab (0.5 mg/kg) Q4W (Part A) | Nemoliozumab (2.0 mg/kg) Q4W (Part A)
Number analyzed (Participants) | 46 | 46 | 45 | 47
change from baseline
  Week 4: number analyzed (Participants) | 43 | 44 | 43 | 46
  Week 4 | -0.2 (0.8) | -0.8 (0.9) | -0.9 (0.9) | -0.6 (0.9)
  Week 8: number analyzed (Participants) | 43 | 44 | 43 | 46
  Week 8 | -0.5 (1.2) | -0.7 (1.0) | -1.0 (1.2) | -0.8 (1.0)
  Week 12: number analyzed (Participants) | 43 | 44 | 43 | 46
  Week 12 | -0.3 (1.0) | -0.7 (1.0) | -1.0 (1.1) | -0.8 (1.1)

7. Secondary Outcome: Changes From Baseline in Static Investigator's Global Assessment (sIGA) (Part A + Part B, ITT Long Population)
Description: as for outcome 6
Time Frame: baseline to Week 12 (Part A), up to Week 64 (Part B)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: change from baseline
Arm/Group | Nemoliozumab (0.1 mg/kg) Q4W (Part A + Part B) | Nemoliozumab (0.5 mg/kg) Q4W (Part A + Part B) | Nemoliozumab (2.0 mg/kg) Q4W (Part A + Part B) | Nemoliozumab (2.0 mg/kg) Q8W (Part A + Part B)
Number analyzed (Participants) | 53 | 54 | 52 | 52
change from baseline
  Week 4: number analyzed (Participants) | 51 | 53 | 50 | 46
  Week 4 | -0.7 (0.9) | -0.8 (0.9) | -0.6 (0.9) | -0.4 (0.8)
  Week 8: number analyzed (Participants) | 48 | 45 | 47 | 42
  Week 8 | -0.8 (1.0) | -1.0 (1.2) | -0.9 (0.9) | -0.5 (0.9)
  Week 12: number analyzed (Participants) | 45 | 46 | 46 | 37
  Week 12 | -0.9 (0.9) | -1.1 (1.1) | -0.9 (1.0) | -0.9 (0.8)
  Week 24: number analyzed (Participants) | 38 | 32 | 37 | 29
  Week 24 | -1.5 (1.1) | -1.7 (1.0) | -1.2 (1.0) | -1.2 (1.1)
  Week 48: number analyzed (Participants) | 32 | 29 | 32 | 20
  Week 48 | -1.7 (1.2) | -1.8 (0.8) | -1.4 (1.2) | -2.0 (1.2)
  Week 60: number analyzed (Participants) | 31 | 28 | 32 | 19
  Week 60 | -1.9 (1.0) | -2.0 (0.9) | -1.7 (1.1) | -1.7 (1.1)
  Week 64: number analyzed (Participants) | 31 | 28 | 29 | 19
  Week 64 | -1.9 (1.1) | -1.9 (0.9) | -1.7 (1.0) | -1.8 (1.3)

8. Secondary Outcome: Changes From Baseline in Body Surface Area (BSA) of Atopic Dermatitis (AD) Involvement (Part A, PP Population)
Description: The total BSA affected by AD was assessed as part of SCORAD. The BSA is a measure of the severity of AD, and it is considered to be severe when the rash with strong inflammation is 10 % or more of the total BSA.
  When the BSA of AD involvement decreases, the change from baseline at each timepoint indicates negative value (i.e. the higher the absolute value is, the more the BSA of AD involvement decreases).
Time Frame: baseline to Week 12 (Part A)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Placebo (Part A) | Nemoliozumab (0.1 mg/kg) Q4W (Part A) | Nemoliozumab (0.5 mg/kg) Q4W (Part A) | Nemoliozumab (2.0 mg/kg) Q4W (Part A)
Number analyzed (Participants) | 46 | 46 | 45 | 47
percentage change from baseline
  Week 4: number analyzed (Participants) | 43 | 44 | 43 | 46
  Week 4 | -7.48 (37.14) | -12.11 (43.69) | -23.49 (40.93) | -18.44 (35.47)
  Week 8: number analyzed (Participants) | 43 | 44 | 43 | 46
  Week 8 | -14.44 (49.29) | -14.90 (45.84) | -27.23 (47.17) | -22.99 (38.58)
  Week 12: number analyzed (Participants) | 43 | 44 | 43 | 46
  Week 12 | -13.29 (49.87) | -17.54 (47.16) | -19.68 (67.49) | -24.36 (41.84)

9. Secondary Outcome: Changes From Baseline in Body Surface Area (BSA) of Atopic Dermatitis (AD) Involvement (Part A + Part B, ITT Long Population)
Description: as for outcome 8
Time Frame: baseline to Week 12 (Part A), up to Week 64 (Part B)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Nemoliozumab (0.1 mg/kg) Q4W (Part A + Part B) | Nemoliozumab (0.5 mg/kg) Q4W (Part A + Part B) | Nemoliozumab (2.0 mg/kg) Q4W (Part A + Part B) | Nemoliozumab (2.0 mg/kg) Q8W (Part A + Part B)
Number analyzed (Participants) | 53 | 54 | 52 | 52
percentage change from baseline
  Week 4: number analyzed (Participants) | 51 | 53 | 50 | 46
  Week 4 | -10.12 (45.56) | -23.28 (38.96) | -17.98 (35.12) | -2.79 (54.12)
  Week 8: number analyzed (Participants) | 47 | 44 | 46 | 42
  Week 8 | -18.08 (45.82) | -29.58 (47.13) | -24.64 (37.49) | -6.66 (59.40)
  Week 12: number analyzed (Participants) | 45 | 46 | 46 | 37
  Week 12 | -24.53 (49.77) | -25.31 (63.43) | -25.91 (44.40) | -18.56 (52.30)
  Week 24: number analyzed (Participants) | 38 | 32 | 37 | 29
  Week 24 | -48.13 (39.07) | -51.41 (44.10) | -40.53 (42.94) | -36.91 (40.99)
  Week 48: number analyzed (Participants) | 32 | 29 | 32 | 20
  Week 48 | -65.21 (32.63) | -69.20 (39.95) | -49.66 (44.18) | -59.97 (50.32)
  Week 60: number analyzed (Participants) | 31 | 28 | 32 | 19
  Week 60 | -60.41 (37.00) | -70.44 (35.81) | -60.99 (48.00) | -58.38 (44.97)
  Week 64: number analyzed (Participants) | 31 | 28 | 29 | 19
  Week 64 | -62.54 (40.92) | -66.01 (36.38) | -63.35 (40.37) | -60.54 (55.96)

ADVERSE EVENTS:
Time Frame: baseline to Week 12 (Part A), up to Week 64 (Part B), Safety Follow-up period
Description: The Investigator is responsible for ensuring that all adverse events are recorded on the Adverse Event eCRF and reported to the Sponsor. For each adverse event recorded on the Adverse Event eCRF, the Investigator will make an assessment of seriousness, severity, and causality.
  Note: The Safety population was used for the analysis. The Safety population included all patients who received at least one dose of Nemoliozumab.
Groups:
- Placebo (Part A): Data from Part A and Safety Follow-up period were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received placebo subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
- Nemoliozumab (0.1 mg/kg) Q4W (Part A): Data from Part A and Safety Follow-up period were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (0.1 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
- Nemoliozumab (0.5 mg/kg) Q4W (Part A): Data from Part A and Safety Follow-up period were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (0.5 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
- Nemoliozumab (2.0 mg/kg) Q4W (Part A): Data from Part A and Safety Follow-up period were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (2.0 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
- Nemoliozumab (2.0 mg/kg) Q8W (Part A): Data from Part A and Safety Follow-up period were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (2.0 mg/kg) subcutaneously every 8 weeks on Day 1 and Week 8.
- Nemoliozumab (0.1 mg/kg) Q4W (Part A + Part B): Data from Part A, Part B and Safety Follow-up period were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (0.1 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
  Active-to-active period (Part B) (up to Week 64):
  Patients in the Nemoliozumab (0.1 mg/kg) Q4W group during Part A continuously used the same regimen of Nemoliozumab in Part B.
- Nemoliozumab (0.5 mg/kg) Q4W (Part A + Part B): Data from Part A, Part B and Safety Follow-up period were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (0.5 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
  Active-to-active period (Part B) (up to Week 64):
  Patients in the Nemoliozumab (0.5 mg/kg) Q4W group during Part A continuously used the same regimen of Nemoliozumab in Part B.
- Nemoliozumab (2.0 mg/kg) Q4W (Part A + Part B): Data from Part A, Part B and Safety Follow-up period were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (2.0 mg/kg) subcutaneously every 4 weeks on Day 1, Week 4 and Week 8.
  Active-to-active period (Part B) (up to Week 64):
  Patients in the Nemoliozumab (2.0 mg/kg) Q4W group during Part A continuously used the same regimen of Nemoliozumab in Part B.
- Nemoliozumab (2.0 mg/kg) Q8W (Part A + Part B): Data from Part A, Part B and Safety Follow-up period were analyzed.
  Placebo-controlled period (Part A) (Day 1 to Week 12):
  Patients randomized to this group received Nemoliozumab (2.0 mg/kg) subcutaneously every 8 weeks on Day 1 and Week 8.
  Active-to-active period (Part B) (up to Week 64):
  Patients in the Nemoliozumab (2.0 mg/kg) Q8W group during Part A continuously used the same regimen of Nemoliozumab in Part B.
Arm/Group | Placebo (Part A) | Nemoliozumab (0.1 mg/kg) Q4W (Part A) | Nemoliozumab (0.5 mg/kg) Q4W (Part A) | Nemoliozumab (2.0 mg/kg) Q4W (Part A) | Nemoliozumab (2.0 mg/kg) Q8W (Part A) | Nemoliozumab (0.1 mg/kg) Q4W (Part A + Part B) | Nemoliozumab (0.5 mg/kg) Q4W (Part A + Part B) | Nemoliozumab (2.0 mg/kg) Q4W (Part A + Part B) | Nemoliozumab (2.0 mg/kg) Q8W (Part A + Part B)
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/53 | 0/54 | 0/52 | 0/52 | 0/53 | 0/54 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/53 | 1/53 | 0/54 | 3/52 | 5/52 | 3/53 | 3/54 | 4/52 | 9/52
Other Adverse Events (participants affected / at risk) | 27/53 | 29/53 | 23/54 | 27/52 | 25/52 | 37/53 | 35/54 | 33/52 | 35/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Part A) (N=53) | Nemoliozumab (0.1 mg/kg) Q4W (Part A) (N=53) | Nemoliozumab (0.5 mg/kg) Q4W (Part A) (N=54) | Nemoliozumab (2.0 mg/kg) Q4W (Part A) (N=52) | Nemoliozumab (2.0 mg/kg) Q8W (Part A) (N=52) | Nemoliozumab (0.1 mg/kg) Q4W (Part A + Part B) (N=53) | Nemoliozumab (0.5 mg/kg) Q4W (Part A + Part B) (N=54) | Nemoliozumab (2.0 mg/kg) Q4W (Part A + Part B) (N=52) | Nemoliozumab (2.0 mg/kg) Q8W (Part A + Part B) (N=52)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 2
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyoderma (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Part A) (N=53) | Nemoliozumab (0.1 mg/kg) Q4W (Part A) (N=53) | Nemoliozumab (0.5 mg/kg) Q4W (Part A) (N=54) | Nemoliozumab (2.0 mg/kg) Q4W (Part A) (N=52) | Nemoliozumab (2.0 mg/kg) Q8W (Part A) (N=52) | Nemoliozumab (0.1 mg/kg) Q4W (Part A + Part B) (N=53) | Nemoliozumab (0.5 mg/kg) Q4W (Part A + Part B) (N=54) | Nemoliozumab (2.0 mg/kg) Q4W (Part A + Part B) (N=52) | Nemoliozumab (2.0 mg/kg) Q8W (Part A + Part B) (N=52)
Nasopharyngitis (Infections and infestations) | 8 | 9 | 6 | 5 | 7 | 15 | 14 | 15 | 12
Upper respiratory tract infection (Infections and infestations) | 6 | 4 | 1 | 4 | 5 | 6 | 3 | 5 | 5
Impetigo (Infections and infestations) | 0 | 4 | 0 | 0 | 0 | 6 | 3 | 0 | 3
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1
Folliculitis (Infections and infestations) | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 7 | 11 | 10 | 9 | 9 | 15 | 12 | 12 | 9
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 1
Oedema peripheral (General disorders) | 0 | 2 | 3 | 5 | 2 | 2 | 3 | 6 | 2
Blood creatine phosphokinase increased (Investigations) | 3 | 2 | 2 | 4 | 3 | 5 | 3 | 9 | 6
Headache (Nervous system disorders) | 0 | 3 | 2 | 3 | 1 | 3 | 6 | 5 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 2 | 1 | 1 | 1 | 3 | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other